CLINICAL TRIAL: NCT00635648
Title: A Non-comparative, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, and Efficacy of Caspofungin Acetate (MK-0991) for the Treatment of Esophageal Candidiasis or Invasive Candidiasis in Chinese Adults
Brief Title: A Study of Caspofungin Acetate (MK0991) for the Treatment of Esophageal Candidiasis or Invasive Candidiasis in Chinese Adults (MK-0991-066)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0991-066; 2008_001
Record Dates: First submitted 2008-02-29; First posted 2008-03-14 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Caspofungin

ARMS (1):
- Caspofungin 50 mg Intravenous (IV) (Experimental)
  Interventions: Drug: caspofungin acetate

INTERVENTIONS:
Drug: caspofungin acetate — Intravenous (IV) caspofungin acetate 50 mg/day. Participants with esophageal candidiasis will be treated for at least 7 days and for at least 72 hours after symptoms resolve for a maximum of 28 days; participants with invasive candidiasis will have a 70 mg loading dose on study day 1 and will be treated for at least 14 days after the last positive culture of Candida from the blood or other normally sterile body site for a maximum of 60 days; these participants should also have improvement in clinical and radiographic signs of disease for at least 48 hours before completion of the study therapy.
  Other Names: MK0991; Cancidas®

SUMMARY:
To evaluate the safety, tolerability, and efficacy of caspofungin for the treatment of esophageal candidiasis and invasive candidiasis to support the registration of caspofungin for these indications in China.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a confirmed diagnosis of esophageal candidiasis or invasive candidiasis for whom IV antifungal therapy is appropriate
* FOR ESOPHAGEAL CANDIDIASIS
* Participant has endoscopic evidence of esophageal candidiasis
* Participant has disease documented by symptoms consistent with esophageal candidiasis and positive stain or wetmount KOH of brushing or biopsy from endoscopy followed by positive culture for Candida or positive histopathologic evidence of Candida infection
* FOR INVASIVE CANDIDIASIS
* Participant has at least 1 positive culture of a Candida species from blood or other normally sterile body site obtained within 96 hours of study entry
* Participant has clinical evidence of infection within 96 hours before study entry
* Temperature >100^◦F (37.8^◦F) on 2 occasions at least 4 hours apart or 1 determination of >101^◦F (38.3^◦F) or clinically significant hypothermia <96.8^◦F (36.0^◦C)
* Systolic blood pressure <90 or ≥30 mm Hg decrease in systolic blood pressure from the participant's normal baseline
* Signs of inflammation at a site infected with Candida

Exclusion Criteria:

* Participant has any of the following abnormal laboratory values: International Normalization Ratio (INR) >1.6 or, if participant is receiving anticoagulants, INR >4.0; bilirubin >5 times the upper limit of normal range;

aspartate aminotransferase (AST, or serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT, or serum glutamic pyruvic transaminase [SGPT]) >5 times the upper limit of normal range

* FOR ESOPHAGEAL CANDIDIASIS
* Participant has Candida disease limited to the oropharynx
* Participant has another cause of esophagitis or has clearly defined ulcers on endoscopy with high likelihood of another non-Candida pathogen
* Participant has other esophageal pathology on endoscopy that is unrelated to acute esophageal candidiasis
* FOR INVASIVE CANDIDIASIS
* Participant has evidence of infection limited to a positive culture for Candida from urine, sputum, catheter tip, indwelling drain, or mucosal or superficial skin surface
* Participant has suspected Candida endocarditis, osteomyelitis, or meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lin DF, Wang JM, Yu YS; Han MZ, Shen ZX, Song SD, Zhang YY. A non-controlled, multicenter, open-label study to evaluate the safety, tolerability, and efficacy of caspofungin acetate for the treatment of invasive candidiasis in Chinese adults . Chin J Infect Chemother. 2014;14(5):379-385. [in Chinese]

RESULTS

PARTICIPANT FLOW:
Groups:
- Caspofungin 50 mg q.d. Intravenous (IV): Three participants with esophageal candidiasis were treated with IV caspofungin 50 mg daily (q.d.) for at least 7 days and for at least 72 hours past the resolution of symptoms for a maximum treatment duration of 28 days.
  After a 70 mg loading dose on Study Day 1, 60 participants with invasive candidiasis were treated with IV caspofungin 50 mg q.d. for at least 14 days after the last positive culture of Candida from the blood or other normally sterile body site for a maximum treatment duration of 60 days.
Period: Overall Study
Arm/Group | Caspofungin 50 mg q.d. Intravenous (IV)
Started | 63
Completed | 26
Not Completed | 37
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 4
Not completed — Rapid progression of baseline disease | 4
Not completed — Use of other antifungal agent needed | 1
Not completed — No improvement after 7-10 days treatment | 4
Not completed — Noncompliance with protocol | 1
Not completed — Other reason | 2

BASELINE CHARACTERISTICS:
Arm/Group | Caspofungin 50 mg q.d. Intravenous (IV)
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug-related Serious Adverse Events
Description: A serious adverse event is one that results in death, disability/incapacity, or hospitalization or is life threatening, a congenital anomaly or birth defect, cancer, an overdose, or otherwise jeopardizes the patient and may require medical intervention.
  A drug-related adverse event is a determination by the investigator physician that the study drug caused the event based on exposure, time course, likely cause, dechallenge (event resolved/improved when drug was discontinued), rechallenge (event resolved/improved when drug was re-introduced), and consistency with the drug profile.
Time Frame: First dose of study drug through 14 days post therapy (maximum 28 days of study drug for esophageal candidiasis, 60 days for invasive candidiasis; mean treatment duration of 14 days)
Measure: Number; unit: Participants
Groups:
- Caspofungin 50 mg q.d. IV: Three participants with esophageal candidiasis were treated with IV caspofungin 50 mg daily (q.d.) for at least 7 days and for at least 72 hours past the resolution of symptoms for a maximum treatment duration of 28 days.
  After a 70 mg loading dose on Study Day 1, 60 participants with invasive candidiasis were treated with IV caspofungin 50 mg q.d. for at least 14 days after the last positive culture of Candida from the blood or other normally sterile body site for a maximum treatment duration of 60 days.
Arm/Group | Caspofungin 50 mg q.d. IV
Number analyzed (Participants) | 63
Participants | 0

2. Secondary Outcome: Number of Participants With One or More Drug-related Adverse Events
Description: A drug-related adverse event is a determination by the investigator physician that the study drug caused the event based on exposure, time course, likely cause, dechallenge (event resolved/improved when drug was discontinued), rechallenge (event resolved/improved when drug was re-introduced), and consistency with the drug profile.
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Caspofungin 50 mg q.d. IV
Number analyzed (Participants) | 63
Participants | 31

3. Secondary Outcome: Number of Participants Who Discontinued Due to a Drug-related Adverse Event
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Caspofungin 50 mg q.d. IV
Number analyzed (Participants) | 63
Participants | 1

4. Secondary Outcome: Number of Participants With Favorable Overall Response for Esophageal Candidiasis or Invasive Candidiasis
Description: Efficacy response for esophageal candidiasis was based on clinical and endoscopic criteria; favorable responses included complete and partial improvement in symptoms and endoscopic lesions.
  Efficacy response for invasive candidiasis was based on microbiological and clinical assessments; favorable responses required both favorable microbiological response (i.e., eradication or presumptive eradication based on symptoms, physical exam, and non-invasive tests) and complete or partial clinical response.
Time Frame: First dose of study drug through up to 60 days of therapy (maximum 28 days of study drug for esophageal candidiasis, 60 days for invasive candidiasis; mean treatment duration of 14 days)
Population: Of the 63 enrolled participants, one participant with invasive candidiasis who withdrew consent before completing the efficacy assessment was not included in the efficacy analyses.
Measure: Number; unit: Participants
Arm/Group | Caspofungin 50 mg q.d. IV
Number analyzed (Participants) | 62
Participants | 36

ADVERSE EVENTS:
Time Frame: First dose of study drug through 14 days post therapy (maximum 28 days of study drug for esophageal candidiasis, 60 days for invasive candidiasis; mean treatment duration of 14 days)
Arm/Group | Caspofungin 50 mg q.d. IV
Serious Adverse Events (participants affected / at risk) | 14/63
Other Adverse Events (participants affected / at risk) | 43/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caspofungin 50 mg q.d. IV (N=63)
Cardiac Failure (Cardiac disorders) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1)
Death (General disorders) | 5 (5)
Renal Failure (Renal and urinary disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Circulatory Collapse (Vascular disorders) | 4 (4)
Hypovolaemic Shock (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caspofungin 50 mg q.d. IV (N=63)
Cardiac Failure (Cardiac disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Oedema (General disorders) | 4 (4)
Pyrexia (General disorders) | 5 (7)
Alanine Aminotransferase Increased (Investigations) | 10 (10)
Aspartate Aminotransferase Increased (Investigations) | 9 (10)
Blood Albumin Decreased (Investigations) | 6 (6)
Blood Bilirubin Increased (Investigations) | 7 (11)
Blood Calcium Decreased (Investigations) | 5 (9)
Blood Creatinine Increased (Investigations) | 7 (8)
Blood Glucose Increased (Investigations) | 4 (4)
Blood Potassium Decreased (Investigations) | 25 (30)
Blood Sodium Decreased (Investigations) | 4 (4)
Blood Urea Increased (Investigations) | 5 (5)
Protein Total Decreased (Investigations) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Platelet Count Decreased (Investigations) | 5 (5)

LIMITATIONS AND CAVEATS:
This was an open-label non-comparative study with a relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Twenty-four months after completion of this study or after publication of the multicenter results, an investigator may publish the results for their study site independently. The sponsor must have the opportunity to review all proposed publications or presentations regarding the study 60 days before submission.